CLINICAL TRIAL: NCT03955861
Title: An Observational Study Evaluating the Utility of Ultrasound Confirmed Enthesitis as a Prognostic Marker for Response to Biologic Therapy in Psoriatic Arthritis
Brief Title: Ultrasound Enthesitis Response in Psoriatic Arthritis
Status: Completed | Type: Observational
Sponsor: Belfast Health and Social Care Trust (Other)
Collaborators: British Medical Association (Other); Psoriasis and Psoriatic Arthritis Alliance (Unknown); Queen's University, Belfast (Other)
Responsible Party: Sponsor
Other Study IDs: 18046MR-SW
Record Dates: First submitted 2019-02-13; First posted 2019-05-20 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-02

CONDITIONS: Psoriatic Arthritis; Psoriasis; Enthesitis
MeSH Terms: conditions — Arthritis, Psoriatic; Psoriasis | interventions — Adalimumab; Certolizumab Pegol; Etanercept; golimumab; secukinumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bloods samples with whole blood/serum/plasma storage for future biomarker analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Biological: adalimumab — Subcutaneous injection
  Other Names: Humira
Biological: Certolizumab — Subcutaneous injection
  Other Names: Cimzia
Biological: Etanercept — Subcutaneous injection
  Other Names: Enbrel
Biological: Golimumab — Subcutaneous injection
  Other Names: Simponi
Biological: Secukinumab — Subcutaneous injection
  Other Names: Cosentyx

SUMMARY:
The aim of this observational study will be to recruit 100 Psoriatic Arthritis (PsA) patients beginning on their biologic therapy and asses, both clinically and with the use of ultrasound (US), how enthesitis responds to biologic treatment.

The decision to start treatment with a biologic therapy will be made by the patients' usual clinical rheumatology team, as part of their standard clinical care. This is independent of the study. Patients in whom treatment with these drugs for their PsA has been recommended will then be invited to participate in this study.They will then be commenced on biologic therapy at doses in line with the Summary of Product characteristics (SPC) for the product and followed up in the hospital outpatient clinic.

Patients will have a full history taken and clinical exam performed prior to commencing on their prescribed biologic. The patient's history, Health Assessment Questionnaire scores and biobanking samples will be taken by the co-investigator. They will also calculate the patients tender and swollen joint score, dactylitis score, skin score, nail score and clinical enthesitis score.They will then have their tender entheseal points scanned as well as those as per the MASEI (Madrid Sonographic Enthesitis Index ) protocol by a single rheumatologist. The rheumatologist will be trained in ultrasound and will perform the scans blinded to this information both at initial consultation and at subsequent reviews.

The patient will then commence their biologic treatment as planned at a separate review as per usual practise with their clinical team.

Follow-up and final assessment at 4 months (±2 weeks) after starting biologic will include the clinical and ultrasound assessments as per the initial review and outlined in the schedule of assessments. They will also have a final blood sample taken at this point.

DETAILED DESCRIPTION:
Objective: This study will aim to clarify, in a cohort of active PsA patients, what is the prevalence of US confirmed enthesitis, what happens to these scores after biologic treatment, does this correlate with clinical scores and can enthesitis then serve as a prognostic tool in predicting response in patients receiving their biologic therapy.

Aims and objectives:

Primary outcome:

-The change in MASEI score at 4 months from baseline assessment.

Study design:

A prospective,assessor-blinded, cohort observational study of biologic-naive patients with PsA receiving biologic treatment as part of standard clinical care.

An observational trial was deemed appropriate to answer the study question and provide real life data to form the basis of future randomised controlled trials.

Duration Participants will be in the study for a maximum of 6 months, with most participants completing the study within 4 months after starting the biologic. The end of the trial will be at the 4 month assessment for the final patient with the locking of the study database.

Study setting The study will be carried out on one site in Musgrave Park Hospital, Belfast. This is an NHS (National Health Service) teaching hospital, part of the Belfast Health and Social Care Trust.

Inclusion and exclusion criteria Inclusion criteria for PsA patients

Patients with PsA will be included if they meet all of the following criteria:

1. Aged ≥ 18 years
2. Fulfil the Classification criteria for PSA (CASPAR criteria)
3. Have not previously had biologic disease modifying treatment for their PsA
4. Are due to commence on subcutaneous TNF (Tumour necrosis Factor) inhibitor or secukinumab as part of their standard clinical care, in line with the product SPC
5. Are able and willing to give informed consent and comply with the requirements of the study protocol NOTE: DMARD therapy will be permitted and used as per standard clinical practice (will be captured in CRF)

Exclusion criteria:

Patients will not be eligible if they meet any of the following criteria:

1. History of or current autoimmune rheumatic disease other than PsA 2. Previously received a biologic therapy for PsA 3. Receiving infliximab (IV TNF inhibitor) 4. Haemoglobin ≤9 g/dl 5. Known Human immunodeficiency Virus (HIV), hepatitis C or B infection 6. Current oral steroids 7. Intramuscular steroids within 6 weeks of baseline (IA steroid injection will be allowed) 8. Pregnancy or breast feeding in line with current prescribing recommendations 9. Prisoners or subjects who are involuntarily incarcerated. 10.Subjects who are compulsorily detained for treatment of either a psychiatric or physical (e.g., infectious disease) illness.

Study procedures:

Initial Patient Approach and consent

The decision to start treatment with subcutaneous biologic therapy will be made by the patients' usual clinical rheumatology team, as part of their standard clinical care. This is independent of the study. Patients in whom treatment with these drugs for their PsA has been recommended will then be invited to participate in this study. The initial approach to potential participants will be by their usual clinical team.

Written informed consent will be obtained from each subject prior to any study-related procedures being performed. Consenting participants will have their baseline study assessment performed whilst on the NHS biologic waiting list. They will then be commenced on biologic therapy, as prescribed and followed up in the hospital outpatient clinic as usual at the 4 months mark.

Initial consultation and blinding

Each group will have a full history taken and clinical exam performed as noted below. They will then have their tender entheseal point scanned as well as those as per the MASEI protocol. The patient's history, HAQ (Health Assessment Questionnaire) scores and biobanking samples will be taken by the co-investigator. The co investigator will be a rheumatology registrar and will then assess skin, joints, nails and enthesitis points and calculate the scores below, all of which are routine tools used in clinical practise. A single rheumatologist trained in US will perform the scans blinded to this information both at initial consultation and at the 4 month review. The co-investigator and participants will not be blinded to the treatment or results, although within the first consultation neither patient or assessor will know what medication the consultant team will ultimately decide to commence the participant on.

Biologic treatment will then be administered as planned by the patient's consultant rheumatologist.

Baseline visit (up to 2 weeks prior to starting biologic):

1. Demographic data and confirmation of inclusion and exclusion criteria
2. Duration of PsA and psoriasis
3. Calculate BMI
4. Social History: Smoking status and alcohol use
5. Family History: Of joint or skin disease
6. Drug history
7. Full clinical exam with height and weight
8. Calculate MDA (Tender joint score 66 Swollen joint score 68 LEI- C or N BSA (Body Surface Area)/ PASI (Psoriasis Area and Severity Index) measurement Patient pain VAS Patient global disease activity VAS HAQ-See attached sheet)
9. Calculate their Spondyloarthritis research consortium of Canada (SPARCC) enthesitis score
10. Calculate their Leeds Enthesitis Score (LEI)
11. Calculate Bath AS disease activity index (BASDAI)
12. Calculate their (Dermatology Life Index score) DLQI score
13. Calculate their Nail Severity Psoriasis Index (NAPSI) score.
14. Calculate their Dactylitis score
15. Calculate their Physician global assessment score
16. Calculate their DAS (Disease Activity Score)-28 score
17. Blood investigations: FBC (Full Blood Count), renal profile, eGFR, inflammatory markers (CRP, ESR) and liver profile will have been taken as part of routine care (Results will be noted)
18. Blood samples for biobanking
19. Imaging Ultrasound Scan entheseal points as per the MASEI score These will include- Six bilateral enthesis locations in each patient, including the proximal plantar fascia, distal Achilles tendon, distal and proximal patellar ligament, distal quadriceps and brachial triceps tendons Modalities to be documented i. Enthesophyte ii. Power Doppler signal iii. Entheseal calcification iv. Erosions v. Entheseal thickness

Ultrasound scan any other entheseal points that are symptomatic, this includes if there is nail changes. Choose one nail bed to US scan to assess for changes.

Sample collection for biobanking At each time point 20ml of additional blood will be collected from each participant each, comprising whole blood (RNA), PBMC (DNA), serum and plasma (for future immunoassays, metabolomics) .This will be placed on ice and transferred securely to Queen University Belfast and spun down and the plasma will be stored at Dr Rooney's Laboratory. All samples will be labelled with a unique patient study participant code and this will be recorded in the database. They will be stored in a freezer at a temperature of at least -20oC. The samples will be anonymised with their unique code and will only be able to be identified by the principal investigator. Analysis will include a targeted or unbiased protein assessment strategy in the form of a mass spectrometry based proteomics platform. Analysis may also include that of genetic variation markers, related to the target pathway of the biologic therapies. This may involve whole genome sequencing.

Patient will then go onto their biologic treatment as planned at a separate appointment with their clinical team where a plan will be put in place for review to assess response to drug as usual at 4 months

Interventions

The decision to commence a patient on a biologic therapy will be made independent of the study protocol by the patient's rheumatology consultant. All study participants will be retained in the trial whenever possible to enable follow-up data collection and prevent missing data.

If a patient has not been able to take their biologic therapy for a period of more than or equal to 6 weeks during the study they will be deemed to not have completed the treatment and will not be included in the final comparative analysis. Each of the biologic medications being used in this study has a marketing authorisation in the UK and is being used in its marketed presentation and packaging bearing the MA number. All medications will be sourced locally by the research site pharmacy in Musgrave Park Hospital at market price as per standard procedure independent of the study and stored and distributed as per usual practices.

Biologic treatment routinely used at Musgrave Park Hospital for PsA are as follows:

1. Etanercept
2. Adalimumab
3. Certolizumab pegol
4. Golimumab
5. Secukinumab

Follow-up and final assessment (4 months ±2 week after starting biologic) Clinical and ultrasound assessments as per the initial review will be carried out without the need to go over exclusion/inclusion criteria, past medical history or family history. An additional PsARC calculation based on response will be made at this point.

A further bio banking sample will be taken at the 4 months mark.

Time plan and Study Centres:

Recruitment will take place during the first 6 months of the study and the study will end 4 months after the recruitment of the last patient. Once the first participant is referred by their consultant they will be put on the biologic waiting list to commence their new medication. This process usually takes 3 months from referral to commencing on their biologic medication. We will assess the participant two weeks prior to this review and then their next review will be at the 4 months mark prior to their second consultant review. The participant involvement will end then.

Sample size Sample size calculation. On reviewing the literature in relation to the MASEI score, the initial paper to highlight its validity as a scanning tool in those with spondyloarthropathy compared with controls was able to demonstrate this with only 25 patients.

In this study 84% of patients demonstrated active disease as defined by a cut off score of 18 and therefore we would expect in a cohort of active PsA patients that the vast majority will demonstrate active disease to allow comparison after biologic treatment. Based then on available data on PsA patients prescribed biologic therapy within the Belfast trust, a sample size of 100 patients was deemed achievable and would allow the primary outcome to be answered.

Assuming 100 patients are recruited split 50/50 between IL (Interleukin)-17 and TNF. Then the study will have 85% power to determine a difference between groups as statistically significant if the difference in MASEI change scores at three months between the two groups is equal to 0.6 standard devia- tions of the change score. This calculation assumes equal variation in the change score in both groups, a significance level of 0.05 and is based on a two-sided hypothesis

Recruitment Patients will first be approached by one of the seven rheumatology consultants, based in Musgrave Park Hospital.If patients are agreeable to hear more information on the research they will be referred to the research team who are based in the Belfast Trust. Initially an email with patient details will be sent to the research team who will telephone the potential participant to discuss the study and verbally explain what the study entails. If the patient is interested in participating in the study they will have an information sheet posted out to their home address. The patient will then attend for their initial consultation and at this point, if they are still happy to proceed with participation, they will be consented for inclusion in the study. Hospital numbers and personal details will be communicated by Trust computers and each patient will be given a unique identifier number once enrolled. During the study the medication the patient is then prescribed by their consultant team will be noted by the co-investigator and/or nurse specialist. The aim will be to recruit at least 2 patients a week with the expected time line to be 12 months to complete recruitment and 18 months at a maximum to complete the final patient assessment.

Data Management Each patient will have a unique study code participant number to make information anonymised. The study will be conducted on NHS property by researchers from the Belfast Health and Social Care Trust and any personal information will be held securely on Trust property and handled in accordance with the provisions of the Data Protection Act 2018. Blood samples will be labelled with the unique study code for each participant prior to storage. These codes will be contained within a master file and will be kept under secure conditions within a locked fill-in cabinet on Belfast Trust property.

Statistical analysis Analysis of MASEI scores will be by independent samples t-tests and Analysis of covariance. Differences between patient groups will be examined by calculating propensity scores, obtained from running a logistic regression analysis with grouping variable as outcome and patient demographic and medical history variables as explanatory. If the propensity analysis is statistically significant the propensity scores will be included in all subsequent analysis of MASEI. Secondary variables will be treated in a similar manner. Firstly the researchers will look as to whether the MDA (5/7) or PsARC (Yes/No) score is achieved at the 4 months assessment. The researchers will also compare the LEI, Dactylitis, 66/68 Tender and swollen score change from baseline to 4 months. Finally the research team will look at the relationship between MASEI score and clinical scores at the 4 months mark to see if there is correlation. The change in US findings at the nail bed will be a descriptive result of any changes noted.

The research team do not envisage any urgent safety measures that will be required a part of this project.

The CI or in exceptional cases the PI will report the urgent safety measure to the Trust Research Office immediately by telephone or within 3 days in written form.

Consent PI (Ashley Elliott) will be taking the written consent of the patient. Once they have been approached to participate by their consultant the participants will receive an information sheet explaining the study. Written consent will be gained at the first consultation.

Declaration of interests There is no financial or other competing interests for the principal investigators for the trial.

ELIGIBILITY:
Inclusion criteria for PsA patients

Patients with PsA will be included if they meet ALL of the following criteria:

1. Aged ≥ 18 years
2. Fulfil the Classification criteria for PSA (CASPAR)
3. Have not previously had biologic disease modifying treatment for their PsA
4. Are due to commence on subcutaneous TNF inhibitor or secukinumab as part of their standard clinical care, in line with SPC for the product prescribed
5. Are able and willing to give informed consent and comply with the requirements of the study protocol NOTE: DMARD therapy will be permitted and used as per standard clinical practice

Exclusion criteria:

Patients will not be eligible if they meet ANY of the following criteria:

1. History of or current autoimmune rheumatic disease other than PsA
2. Previously received a biologic therapy for PsA
3. Receiving infliximab (IV TNF inhibitor)
4. Haemoglobin ≤9 g/dl
5. Known HUMAN immunodeficiency Virus (HIV), hepatitis C or B infection
6. Current oral steroids
7. Intramuscular steroids within 6 weeks of baseline (IA steroid injection will be allowed) assessment
8. Pregnancy or breast feeding
9. Subjects who are compulsorily detained for treatment of either a psychiatric or physical (e.g., infectious disease) illness. -

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Psoriatic Arthritis patients with active disease who are naive to biologic therapy
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2019-02-14 (Actual); Primary Completion 2021-07-17 (Actual); Study Completion 2021-07-17 (Actual)

PRIMARY OUTCOMES:
The change in Madrid enthesitis ultrasound index (MASEI) score | 4 months
  Ultrasound enthesitis response score. This is a validated tool for assessing enthesitis in spondyloarthropathy. It assess both chronic a active features of enthesitis at the knee, plantar fascia, achilles tendon and triceps tendon. A total score of 136 can be achieved.

SECONDARY OUTCOMES:
The change in Minimal Disease Activity (MDA) response from baseline assessment | 4 months
  Composite clinical score for Psoriatic Arthritis. To be classified as MDA you need to achieve a score of at least 5/7 in the following parameters.
  * Swollen Joint count of ≤ 1 of 66
  * Tender joint score of ≤ 1 out of 68
  * Either a PASI (Psoriasis Area Severity Index) skin score ≤ 15 or a Body Surface Score (BSA) of ≤ 3%
  * Patient Pain Visual Analogue Score (VAS) of ≤ 15
  * Patient Global Disease Activity VAS of ≤ 20
  * HAQ ≤ 0.5
  * Tender Entheseal score of ≤1out of 6 as per the Leeds Enthesitis score
The change in Leeds Enthesitis Index (LEI) score from baseline assessment | 4 months
  Enthesitis clinical score that gives a score out of 6 based on clinical exam of entheseal sites at
  * Both Lateral Epicondyle of the Humerus
  * Both Medial Condyle of the Femur
  * Both Achilles insertion
The change in Dactylitis score from baseline assessment | 4 months
  Dactylitis is the uniform swelling of a whole digit such that the joints cannot be identified. Tenderness when examining dactylitis should be recorded. One dactylitic digit = one swollen joint and score is out of 20 for all five digits.
The change in 66/68 tender and swollen joint counts from baseline assessment | 4 months
  Validated tool to assess 68 sites for tender joints and 66 sites for swollen joints above and below the waist in Psoriatic Arthritis
The change in Psoriatic Arthritis Response Criteria (PsARC) response from baseline assessment | 4 months
  Composite disease activity score in Psoriatic Arthritis
  The PsARC is defined as improvement in at least two of the following 4 criteria (one of which must be tender joint or swollen joint score) with no worsening of any criteria:
  20% or more improvement in physician global assessment of disease activity 20% or more improvement in patient global assessment of disease activity 30% or more improvement in tender joint count 30% or more improvement in swollen joint count
Assess change in Ultrasound (US) findings at nail bed | 4 months
  Nail bed semi quantitative score changes looking at nail bed matrix thickness, nail plate morphology, colour doppler signal and nail bed thickness
Relationship of baseline MASEI score to the clinical outcomes at baseline | 4 months
  A regression analysis will be a carried out on the improvement in participant ultrasound enthesitis scores at 4 months with relation to clinical outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Madeleine Rooney, MD, Study Director — Queens University, Belfast
Locations (1):
- Musgrave Park Hospital, Belfast, Antrim, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Elliott A, Pendleton A, Wright G, Rooney M. The relationship between the nail and systemic enthesitis in psoriatic arthritis. Rheumatol Adv Pract. 2021 Nov 19;5(3):rkab088. doi: 10.1093/rap/rkab088. eCollection 2021. PMID 34888436